CLINICAL TRIAL: NCT04028544
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Study of Qishenyiqi Drop Pills in Improving the Prognosis of Heart Failure Patients With Reduced Ejection Infarction
Brief Title: The Study of Qishenyiqi Drop Pills in Improving the Prognosis of Heart Failure Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Collaborators: Tianjin Tasly Pharmaceutical Co., Ltd (Industry)
Responsible Party: Principal Investigator, Jian Zhang, the director of the heart failure center, Chinese Academy of Medical Sciences, Fuwai Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2015-ZX55
Record Dates: First submitted 2019-06-13; First posted 2019-07-22 (Actual); Last update posted 2019-07-22 (Actual); Status verified 2019-06

CONDITIONS: Heart Failure
Keywords: heart failure; traditional Chinese medicine; prognosis; Qishenyiqi
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The Treatment Group (Experimental): standard treatment + Qishenyiqi dropping pills (QSYQ) (oral use, 1 bag each time, three times a day)
  Interventions: Drug: Qishenyiqi dropping pills
- The Control Group (Placebo Comparator): standard treatment + placebo (oral use, 1 bag each time, three times a day).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Qishenyiqi dropping pills — on the basis of standard treatment, adding QSYQ dropping pills 1 bag each time, 3 times a day
  Other Names: QSYQ
  Arms: The Treatment Group
Drug: Placebo — on the basis of standard treatment, adding placebo 1 bag each time, 3 times a day
  Other Names: Placebo for QSYQ
  Arms: The Control Group

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled study including patients with ejection fraction decreased heart failure under standardized treatment, to evaluate QiShenYiQi (QSYQ) dropping pill's curative effect in reducing cardiovascular death and heart failure rehospitalization compared with placebo.

DETAILED DESCRIPTION:
This is a prospective, large-scale samples, randomized, double-blind, placebo parallel-controlled, multicenter study to evaluate QSYQ's curative effect in reducing cardiovascular death and heart failure rehospitalization in patients with ejection fraction decreased heart failure（LVEF≤40%）under standardized treatment. The results will provide clinical evidence for combined treatment of traditional Chinese medicine and western medicine in ejection fraction decreased heart failure.

There are two treatment groups in the study, which are the treatment group with standard treatment + QSYS (oral use, 1 bag each time, three times a day) , and the control group with standard treatment + placebo (oral use, 1 bag each time, three times a day) .

The subjects are patients with ejection fraction decreased (≤40%) heart failure (NYHA II-IV). The sample size is 5380. For the primary end event, type I error is bilateral 0.05, and POWER was 0.8. The CV death and the HF readmission rate in the trial control group is 15%, and 12.7% in the experimental group. The trial cycle is about 3 years. A total of 4373 subjects will be assigned to the experimental group and the control group at a proportion of 1:1. The primary endpoint was expected to be 1211 cases. Taking into account the annual rate of lost to follow-up is about 18%, the final sample cases is 5380. During the treatment period and extends to at most 2weeks after treatment, patients will get examination including interviews (direct inquiries about the occurrence of adverse events and the situation of taking drugs), physical examination, body weight and the ECG. Laboratory parameters to evaluate clinical safety, such as routine blood, serum creatinine and urea nitrogen, electrolyte (serum potassium, sodium and chloride) and liver enzymes will be taken regularly. Researchers need to record and evaluate any occurrence of adverse events (AE) or serious adverse event (SAE) and its relevance to study medicine.

The primary endpoint is to evaluate whether QSYQ can reduce cardiovascular death and heart failure rehospitalization in chronic heart failure patients with reduced ejection infarction (HFREF) compared with placebo.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand the requirements of the study and willingness to provide written informed consent.
* Male or female subjects aged ≥ 18 years
* Patients with ejection fraction decreased heart failure (NYHA II-IV, Echocardiography with Simpson method within four weeks and NT-proBNP within two weeks before random) （1）35%≤LVEF≤40% ; NT-proBNP≥900pg/ml, patients with renal dysfunction (glomerular filtration rate <60 ml/min/1.73m2）or atrial fibrillation, the NT-proBNP should be ≥1200 pg/ml； （2）LVEF<35% (Simpson method); NT-proBNP≥600pg/ml, patients with renal dysfunction (glomerular filtration rate <60 ml/min/1.73m2）or atrial fibrillation, the NT-proBNP should be ≥900 pg/ml.
* A history of hospitalization or emergency treatment for heart failure in the past two years and a diagnosis of heart failure at least one month ago
* The use of medications in line with the recommendation of China heart failure treatment guidelines for at least 4 weeks. (Please confirm that all the following conditions must be met) : Including a ACEI or ARB, and a beta- blocker, unless contraindicated or not tolerated. The doses should reach the target dose recommended by the guideline or the maximum dose that the patient can tolerate, and the doses should not be changed within one months prior to screening and randomization (patients not take such drugs according to the guidelines, should be recorded).

Exclusion Criteria:

* Acute decompensated HF with hemodynamic instability, mechanical hemodynamic support or invasive mechanical ventilation within 14 days of randomization, using intravenous positive inotropic drugs, vasoactive drugs and intravenous diuretics within 7 days before randomization.
* Poorly controlled hypertension, defined as resting systolic blood pressure≥180mmHg and /or diastolic blood pressure ≥110mmHg assessed on two separate occasions prior to randomization.
* Liver transaminase (ALT or AST), bilirubin more than 3 times the upper limit of normal not caused by heart failure, glomerular filtration rate<15ml/min/1.73m2.
* Hemoglobin concentration ≤ 9.0g/dl and/or have blood system disease.
* Valvular heart disease, congenital heart disease without surgery.
* Cardiac shock.
* Hypertrophic obstructive cardiomyopathy, restrictive cardiomyopathy, other secondary and invasive cardiomyopathy.
* Active myocarditis.
* Constrictive pericarditis, other pericardial diseases.
* Syncope within 3 months.
* Symptomatic bradycardia or II or III degrees heart block without a pacemaker.
* Ventricular arrhythmias affecting hemodynamics.
* Cardiac resynchronization therapy implanted pacemaker (CRT-P) or cardiac resynchronization therapy defibrillators (CRT-D) within 6 months, or upgrade the existing conventional pacemaker or implantable implantable defibrillator (ICD) to the CRT device, or have the intention to implant similar devices.
* Occurred within 3 months: acute coronary syndrome, stroke, transient ischemic attack; Heart, carotid artery or other large vascular surgery; Percutaneous coronary intervention (PCI) or carotid artery angioplasty, CABG or other cardiac surgery.
* Major surgery within 6 months prior to randomization.
* Has a history of heart transplantation or are waiting for transplants or using left ventricular assist device (LVAD) or have intention to heart transplant (waiting for transplants) or implant the VAD.
* Severe chronic obstructive pulmonary disease, pulmonary heart disease, sever pulmonary vascular disease, pulmonary hypertension caused by autoimmune disease, any type of severe pulmonary hypertension.
* History of major organ transplant (such as lung, liver, heart, bone marrow, kidney).
* Patients with serious primary diseases of liver, kidney, hematopoietic system, nervous system, endocrine system, and patients with cancer or mental illness.
* Life expectancy is less than 1 year.
* Known allergy to any study drug.
* Participants in other clinical studies within 1 month.
* Patients who are taking Chinese medicine and proprietary Chinese medicine with similar ingredients of QSYQ.
* Women who have developed pregnancy (pregnancy test positive) or during lactation; women of childbearing age have not taken adequate contraceptive measures.
* According to the researchers, patients could not complete the study or fail to comply with the requirements of the study (due to management or other reasons).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5380 (Estimated)
Dates: Start 2019-03-26 (Actual); Primary Completion 2020-09 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Time to the occurrence of cardiovascular (CV) death or heart failure (HF) re-hospitalization. | up to 30 months
  Compared with placebo, whether QSYQ prolong the occurrence of CV death or HF re-hospitalization of patients with chronic heart failure with lower ejection fraction (HFrEF). The treatment arm with the delayed events happening will be deemed as having a successful response.

SECONDARY OUTCOMES:
Time to the occurrence of all-cause death. | up to 30 months
  Compared with placebo, whether QSYQ prolong the occurrence of all-cause death of patients with HFrEF. The treatment arm with the delayed events happening will be deemed as having a successful response.
Time to the occurrence of all-cause death or HF re-hospitalization. | up to 30 months
  Compared with placebo, whether QSYQ prolong the occurrence of all-cause death or HF re-hospitalization of patients with HFrEF. The treatment arm with the delayed events happening will be deemed as having a successful response.
Time to the occurrence of CV death. | up to 30 months
  Compared with placebo, whether QSYQ prolong the occurrence of CV death of patients with HFrEF. The treatment arm with the delayed events happening will be deemed as having a successful response.
Time to the occurrence of total HF re-hospitalization. | up to 30 months
  Compared with placebo, whether QSYQ prolong the occurrence of total HF re-hospitalization of patients with HFrEF. The treatment arm with the delayed events happening will be deemed as having a successful response.
Time to the occurrence of composite endpoint. | up to 30 months
  Compared with placebo, whether QSYQ prolong the occurrence of composite endpoint (CV death, hospitalization for deteriorating heart failure, hospitalization for nonfatal myocardial infarction, and hospitalization for nonfatal stroke) of patients with HFrEF. The treatment arm with the delayed events happening will be deemed as having a successful response.
Time to the first occurrence of HF hospitalization. | up to 30 months
  Compared with placebo, whether QSYQ prolong the first occurrence of HF hospitalization of patients with HFrEF. The treatment arm with the delayed events happening will be deemed as having a successful response.
Change from baseline to week 48 for the Kansas City Cardiomyopathy Questionnaire (KCCQ) clinical summary score. | from baseline to week 48
  Compared with placebo, whether QSYQ improve the KCCQ score of patients with HFrEF at the 48th week. KCCQ is a 23-item, self-administered instrument that quantifies physical function, symptoms (frequency, severity and recent change), social function, self-efficacy and knowledge, and quality of life. KCCQ clinical summary score is a composite assessment of physical limitations and total symptom scores. Scores are transformed to a range of 0-100, in which higher scores reflect better health status.
Change from baseline to week 48 for the 6 minutes walking distance. | from baseline to week 48
  Compared with placebo, whether QSYQ improve the 6 minutes walking distance of patients with HFrEF at the 48th week.

OTHER OUTCOMES:
Time to the occurrence of HF death. | up to 30 months
  Compared with placebo, whether QSYQ prolong the occurrence of HF death of patients with HFrEF. The treatment arm with the delayed events happening will be deemed as having a successful response.
Time to the occurrence of total re-hospitalization for nonfatal myocardial infarction and nonfatal stroke. | up to 30 months
  Compared with placebo, whether QSYQ prolong the occurrence of total re-hospitalization for nonfatal myocardial infarction and nonfatal stroke of patients with HFrEF. The treatment arm with the delayed events happening will be deemed as having a successful response.
The improvement of Kansas City Cardiomyopathy Questionnaire (KCCQ) score and sub-domain score. | up to 30 months
  Compared with placebo, whether QSYQ increases KCCQ score and each sub-domain score, to evaluate whether QSYQ has better effectiveness in improving health-related quality of life. Values for the domains range from 0 to 100 with higher scores indicating lower symptom burden and better quality of life. Subdomains include physical limitation, symptoms, quality of life, social limitation, symptom stability, and self-efficacy-the first 4 are combined into an overall summary scale.
Level of NT-proBNP in patients with HFrEF | from baseline to week 24 and week 48
  Compared with placebo, whether QSYQ decrease the NT-proBNP level in patients with HFrEF at the 24th week and the 48th week.
Value of LVEF in patients with HFrEF | from baseline to week 48
  Compared with placebo, whether QSYQ improve the LVEF in patients with HFrEF at the 48th week.
Level of BNP in patients with HFrEF. | from baseline to week 48
  Compared with placebo, whether QSYQ decreases the level of BNP in patients with HFrEF at the 48th week.
Value of clinical comprehensive score in patients with HFrEF. | from baseline to week 48
  Compared with placebo, whether QSYQ improves the clinical comprehensive score in patients with HFrEF at the 48th week.
  Clinical comprehensive score is a 7-scale from the best improvement to the worst deterioration assessed by researchers according to the three components: change of NYHA class level, patients' global self-assessment (assessed by patients themselves according to a 7-scale, from the best improvement to the worst deterioration) and occurence of major adverse event (defined as cardiovascular mortality and heart failure hospitalization).
Effectiveness in reducing medical cost and increasing Quality-adjusted life year （QALYs）in patients with HFrEF. | up to 30 months
  Compared with placebo, whether QSYQ reduces the medical cost and increases the QALYs in patients with HFrEF at the end of treatment, to evaluate the pharmacoeconomic effect.

CONTACTS AND LOCATIONS:
Overall Officials: Jian Zhang, MD, Study Chair — Heart Failure Center, Fuwai Hospital
Locations (1):
- Fuwai Hospital, Beijing, Beijing Municipality, China